CLINICAL TRIAL: NCT05169008
Title: A Multicenter, Randomized, and Open-label Clinical Trial to Evaluate the Safety and Immunogenicity of Intramuscular and Inhaled COVID-19 Vaccine in Children Aged 6-12 Years and Adolescents Aged 13-17 Years Who Have Been Immunized With Two Doses of CoronaVac
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Ad5-nCoV and Ad5-nCoV-IH in CoronaVac Immunized Children and Adolescents
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty recruiting subjects, so the study was terminated.
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Beijing Institute of Biotechnology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CS-CTP-AD5NCOV-PDⅢ
Record Dates: First submitted 2021-12-10; First posted 2021-12-23 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: COVID-19 Vaccine; Inhalation; Ad5; Safety; Immunogenicity; Children; Adolescents
MeSH Terms: conditions — COVID-19; Respiratory Aspiration; Alzheimer Disease 5

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccine Group (Experimental): 1000 participants，500 children aged 6-12 years and 500 adolescents aged 13-17 years, Ad5-nCoV or Ad5-nCoV-IH, ≥90 days after two doses of CoronaVac. Intramuscular injection or nebulized inhalation.
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector); Biological: Recombinant COVID-19 vaccine (adenovirus type 5 vector) for Inhalation (Ad5-nCoV-IH)

INTERVENTIONS:
Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) — Intramuscular injection
Biological: Recombinant COVID-19 vaccine (adenovirus type 5 vector) for Inhalation (Ad5-nCoV-IH) — Nebulized inhalation through the mouth

SUMMARY:
This is a multicenter, randomized, and open-label study to evaluate the immune responses and safety profiles of children aged 6-12 years and adolescents aged 13-17 years receiving Ad5-nCoV (intramuscular injection) or Ad5-nCoV-IH (nebulized inhalation) ≥ 90 days after receiving two doses of CoronaVac.

DETAILED DESCRIPTION:
A total of 1000 participants will be equally divided into the two study groups, children of 6-12 years and adolescents of 13-17 years. In each age group, they will have an equal chance to received either one dose of Ad5-nCoV (intramuscular injection) or Ad5-nCoV-IH (nebulized inhalation). The enrollment of the children group will start after the safety profiles in 7 days post-vaccination of the adolescent group have been deemed acceptable. Investigators should try to balance the age and sex of the participants during enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-12 years and adolescents aged 13-17 years at the time of randomization.
2. Have received a complete two dose schedule of CoronaVac for ≥ 90 days.
3. Obtain written informed assent from participants and consent from parents, guardians or legal representatives.
4. Subjects are eligible for immunization of this product as evaluated by investigators after medical history examination, physical examination and clinical judgment of health.

Exclusion Criteria:

1. Have a history of seizures, epilepsy, encephalopathy, psychosis.
2. History of anaphylaxis to any vaccine component.
3. Positive urine pregnancy test result, pregnant, lactation women. Female had menarche must conduct the urine pregnancy test.
4. Congenital or acquired angioedema/neuroedema .
5. Medical history of Guillain-Barré syndrome.
6. Have had asthma attacks within 2 years.
7. Have severe nasal or oral diseases, such as rhinitis (sinusitis), allergic rhinitis, oral ulcer, throat swelling, etc.
8. Asplenia or functional absence of spleen.
9. Bleeding disorder (e.g. protein S or factor deficiency, coagulopathy or platelet disorder).
10. Any confirmed or suspected immunosuppressive or immunodeficient state; received immunosuppressive therapy, cytotoxic therapy, or chronic corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis and surface corticosteroid therapy for acute non-complicated dermatitis) within the past 6 months.
11. Have chronic systematic infection or chronic pulmonary disease
12. Administration of immunoglobulins and/or any blood products within three months prior to the planned administration of the vaccine candidate.
13. Receiving anti-tuberculosis or cancer treatment.
14. History of COVID-19 disease.
15. Have a positive result at the examination of rapid SARS-CoV-2 antibody assay (S-RBD IgG) before vaccination.
16. Have received COVID vaccines other than CoronaVac.
17. Received or plan to receive any non-COVID vaccines (licensed or investigational), within 14 days before and after study vaccination.
18. Current diagnosis of or treatment for cancer, e.g. leukemia.
19. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, and affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Incidence of SAE | Day 0 to 12 months post IM or IH
  Evaluate the incidence of severe adverse events (SAE)
Immunogenicity of S-RBD IgG antibody | 28 days post IM or IH
  GMC of S-RBD IgG antibody by Elisa post vaccination

SECONDARY OUTCOMES:
Incidence of Adverse Reactions (ARs) | Within 14 days post IM or IH
  Incidence of solicited adverse reactions (ARs)
The incidence of AR and AE | Within 28 days post IM or IH
  Incidence of AR and AE within 28 days
Immunogenicity of S-RBD IgG antibody | 14 days post IM or IH
  GMC of S-RBD IgG antibody post vaccination by ELISA
Immunogenicity of S-RBD IgG antibody | 14 and 28 days post IM or IH
  Seroconversion rate of S-RBD IgG antibody post vaccination by ELISA
Immunogenicity of S-RBD IgG antibody | 14 and 28 days post IM or IH
  GMI of S-RBD IgG antibody post vaccination by ELISA
Immunogenicity of S-RBD IgG antibody | 14 and 28 days post IM or IH
  GMT of pseudo-virus neutralizing antibody by ELISA
Immunogenicity of S-RBD IgG antibody | 14 and 28 days post IM or IH
  GMI of pseudo-virus neutralizing antibody by ELISA
Immunogenicity of S-RBD IgG antibody | 14 and 28 days post IM or IH
  Seroconversion rate of pseudo-virus neutralizing antibody by ELISA

OTHER OUTCOMES:
Efficacy of booster vaccination | Up to 12 months post IM or IH
  The number of all COVID-19 cases after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Stephania Passalacqua, Principal Investigator — Hospital Base de Osorno, Chile
Locations (2):
- Chile (2):
  - Hospital Base de Osorno, Osorno, Los Lagos Region
  - Hospital Carlos van Buren, Valparaíso, Región de Valparaíso

IPD SHARING:
Plan to Share IPD: No